CLINICAL TRIAL: NCT01540500
Title: An Open-label, Single-sequence Study in Healthy Subjects to Evaluate the Single-dose Pharmacokinetics of Tasimelteon Alone and in Combination With a CYP1A2 Inhibitor, Fluvoxamine
Brief Title: Pharmacokinetics of Tasimelteon Alone and in Combination With CYP1A2 Inhibitor, Fluvoxamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1111
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — tasimelteon; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Steady State PK Group (Experimental)
  Interventions: Drug: Tasimelteon; Drug: Fluvoxamine

INTERVENTIONS:
Drug: Tasimelteon — 5.66 mg dose on Day 1 and Day 8
  Other Names: VEC-162; BMS-214778
Drug: Fluvoxamine — 50 mg Dose on Days 2-8

SUMMARY:
The purpose of this research study is to evaluate whether administration of a CYP1A2 inhibitor affects the single-dose pharmacokinetics of tasimelteon and its metabolites. The safety and tolerability of tasimelteon will also be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 18 - 55 years, inclusive;
2. Non-smokers [abstinence from smoking for at least 6 months before the screening visit] and test negative for cotinine at screening and baseline;
3. Subjects with Body Mass Index (BMI) of ≥18 and ≤35 kg/m2 (BMI = weight (kg)/ [height (m)]2);
4. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing and females must have a negative pregnancy test at the screening and baseline visits;
5. Note 1: Acceptable methods of birth control include any one of the following: abstinence, vasectomized sexual partner, hormonal methods (i.e. pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam.
6. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   * Body temperature between 35.0-37.5 °C;
   * Systolic blood pressure between 90-150 mmHg;
   * Diastolic blood pressure between 50-95 mmHg;
   * Pulse rate between 50-100 bpm.
7. Ability and acceptance to provide written informed consent;
8. Willing and able to comply with study requirements and restrictions;
9. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests.

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse or evidence of such abuse as indicated by the laboratory assays conducted during the Screening Visit or at Baseline;
2. Any major surgery within three months of Baseline or any minor surgery within one month;
3. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction judged by the Investigator to be clinically significant;
4. Subjects who are currently considered a suicide risk, any subject who has ever made a suicide attempt, or those who are currently demonstrating active (within the last year) suicidal ideation as deemed by the Columbia Suicide Severity Rating Scale (C-SSRS);
5. Any condition requiring the regular use of medication except those listed on Section 8.2;
6. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of baseline;
7. Anyone who has taken a melatonin preparation chronically within the past two months prior to Day 1;
8. Donation or loss of 400 mL or more of blood within two months prior to the Baseline Visit;
9. Significant illness within the two weeks prior to Baseline;
10. A known intolerance or hypersensitivity to fluvoxamine, tasimelteon or drugs similar to tasimelteon (including melatonin) or fluvoxamine;
11. Pregnant or lactating females;
12. History of liver disease and/or positive for one or more of the following serological results:

    * A positive hepatitis C antibody test (anti-HCV)
    * A positive hepatitis B surface antigen (HBsAg)
    * A positive HIV test result
13. Exposure (within 2 weeks of the Baseline Visit) of any over-the-counter medications including dietary supplements and/or herbal remedies, except those listed on Section 8.2;
14. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 days preceding the Screening visit;
15. Participation in a previous BMS-214778/VEC-162 trial;
16. Use of any food or beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats for at least 2 weeks before the Baseline Visit until the end of the study;
17. Inability to be venipunctured and/or tolerate venous access;
18. Subjects who are unable to read or speak English;
19. Any other sound medical reason as determined by the clinical Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Tasimelteon pharmacokinetic parameters (AUC, Cmax, Tmax) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12 and 24 hours post-dose.

SECONDARY OUTCOMES:
Safety and tolerability as measured by spontaneous reporting of AEs, and clinically significant changes in laboratory parameters, ECG parameters, and vital signs | Days 1-9
The Columbia Suicide Severity Rating Scale will be used to assess suicidal behavior and ideation. | Screening, Day -1 (baseline), and Day 9 (end of study)
Pharmacokinetic parameters (AUC, Cmax, Tmax) of tasimelteon metabolites M9, M11, M12, M13, and M14 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12 and 24 hours post-dose.
Fluvoxamine pharmacokinetic parameters (AUC, Cmax, Tmax) | Pre-dose, 1, 3, 4, 6, 8, 12, and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States